CLINICAL TRIAL: NCT00525694
Title: Determination of Clinically Significant Carbohydrates Added to Zero Calorie Drink Products
Brief Title: Zero Calorie Drink Products
Acronym: GGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CCC27009
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): glucose tolerance test solution
  Interventions: Other: Glucose tolerance test; Other: glucose tolerance test solution
- 2 (Other): Diet Coke
  Interventions: Other: Diet Coke
- 3. (Other): Coke Zero
  Interventions: Other: Coke Zero

INTERVENTIONS:
Other: Glucose tolerance test — 10 ounces glucose tolerance test solution
  Arms: 1
Other: glucose tolerance test solution — 75 grams glucose load
  Arms: 1
Other: Diet Coke — 10 ounces of Diet Coke
  Arms: 2
Other: Coke Zero — 10 ounces of Coke Zero
  Arms: 3.

SUMMARY:
This will be a clinical test to determine if any carbohydrate or a gluconeogenic precursor added to a zero calorie product might be important to consider in the management of obesity, metabolic syndrome and diabetes mellitus. This research trial will evaluate the effect of three different solutions on blood glucose level. One solution is plain water, the second a standard high glucose (sugar) solution used typically in diabetes testing, and the third a low calorie drink (Zero Coke). Based on a prior study evaluating a diet for effective weight loss, we observed that patients who drank large volumes of diet soda did not lose weight as readily as those who did not drink diet soda. Therefore, we propose to examine the actual effect of one diet soda (Zero Coke) on the body's glucose level and compare it to water and a high glucose solution. All participants in this study must have 3 Glucose tolerance evaluations - one with each solution: water, high glucose, and Zero Coke.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* asymptomatic individuals for diabetes and pre-diabetes,
* especially for people at high risk of developing diabetes,
* such as those with a family history of diabetes,
* those who are overweight,
* and those who are more than 40 to 45 years old

Exclusion Criteria:

* Patients with chronic illnesses, especially diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
to determine if any carbohydrate or a gluconeogenic precursor added to a zero calorie product might be important to consider in the management of obesity, metabolic syndrome and diabetes mellitus. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: James Hays, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States